CLINICAL TRIAL: NCT02512731
Title: Intraoperative Fluid Therapy for Deceased Donor Renal Transplantation
Acronym: EDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: REB 11-0055-A
Record Dates: First submitted 2015-04-23; First posted 2015-07-31 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal directed fluid therapy using esophageal doppler monitor (Active Comparator): The esophageal doppler monitor directs the fluid therapy.
  Interventions: Device: Esophageal Doppler Monitor
- Fluid therapy using standard management (No Intervention): The esophageal doppler monitor is in place however blinded to the healthcare providers, fluid management is as per standard clinical practice.

INTERVENTIONS:
Device: Esophageal Doppler Monitor — Esophageal doppler monitoring (EDM) is a minimally invasive means of continuously measuring the cardiac output from the pattern of blood flow in the descending thoracic aorta.
  Arms: Goal directed fluid therapy using esophageal doppler monitor

SUMMARY:
Delayed graft function (DGF) is defined as requirement for dialysis in the first week following kidney transplantation. DGF is a common complication occurring in 39% of the deceased donor renal transplants at the investigators' institution with significant cost and outcome implications. The 3 major risk factors for DGF are donor graft characteristics, recipient factors and perioperative management. The most easily modifiable of these factors is perioperative management, in particular intraoperative fluid therapy. The investigators propose to compare the amount of fluid administered using the current standard of care with the fluid administered when optimizing the cardiac output (CO) using Esophageal Doppler Monitoring (EDM) to guide fluid therapy. EDM measures blood flow in the descending aorta, optimizing stroke volume (SV) and cardiac output (CO) by indicating when fluid administration fails to produce an increase in CO.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* signed informed consent
* listed for deceased donor transplantation.

Exclusion Criteria:

* esophageal surgery or cancer
* esophageal stricture, varices or diverticulum
* upper airway surgery
* coarctation of the aorta
* significant valvular heart disease
* clinically significant cardiac arrhythmias
* patient randomized to other trials with an outcome variable of delayed graft function or early graft function will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The volume of crystalloid solutions administered intraoperatively. | Start of Anesthesia until the doppler is removed at the end of surgery, approximately 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Corbella D, Toppin PJ, Ghanekar A, Ayach N, Schiff J, Van Rensburg A, McCluskey SA. Cardiac output-based fluid optimization for kidney transplant recipients: a proof-of-concept trial. Can J Anaesth. 2018 Aug;65(8):873-883. doi: 10.1007/s12630-018-1118-y. Epub 2018 Apr 10. PMID 29637407